CLINICAL TRIAL: NCT02551731
Title: A Phase 2 Study to Assess the Efficacy and Safety of Cannabidiol Oral Solution for the Treatment of Refractory Infantile Spasms
Brief Title: Cannabidiol Oral Solution for Treatment of Refractory Infantile Spasms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor elected not to continue with study
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS011-15-054
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Spasms, Infantile
MeSH Terms: conditions — Spasms, Infantile | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol Oral Solution: 20 or 40 mg/kg/day BID (Experimental): The dose of Cannabidiol Oral Solution will begin at 20 mg/kg/day [10 mg/kg twice per day (BID)], will be adjusted at any time if the investigator feels the safety or well-being of the participant is at risk, and will be titrated up or down according to protocol-stipulated parameters and at the investigator's discretion after Day 14 to enhance efficacy. Dose will not exceed 40 mg/kg/day.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — 20 or 40 mg/kg/day BID

SUMMARY:
Infantile Spasms (IS) is a diagnosis described as a fairly rare and terrible form of epilepsy that usually strikes children in the first year of life. There is a great need for safe and effective therapies in the treatment of IS. This need is even more important for infants and toddlers still sick after being treated with medicine that is already available.

This is a multi-center study to evaluate the efficacy and safety of Cannabidiol Oral Solution (CBD) in the treatment of children aged 6 months through 36 months with a diagnosis of infantile spasms who have not responded to first line therapies.

The overall study duration is expected to be 64 weeks for those subjects who respond to CBD treatment. The maximum possible study duration for each patient is approximately 64 weeks, however a subject will be deemed to have completed the study after 58 weeks.

DETAILED DESCRIPTION:
A protocol amendment in May 2016 created two parts to this trial: Part A (the extended treatment period) and Part B (the safety treatment period), whose objectives are as follows:

Primary Part A: To evaluate the efficacy of Cannabidiol Oral Solution in treating refractory infantile spasms (IS).

Secondary:

Part A:

* To evaluate the safety of Cannabidiol Oral Solution in treating refractory infantile spasms.

Part B:

* To assess the long-term safety of Cannabidiol Oral Solution as an adjunctive treatment for subjects with Infantile Spasms (IS)
* To establish the continued efficacy of Cannabidiol Oral Solution in maintaining seizure control in subjects with IS
* To assess the global status of subjects taking Cannabidiol Oral Solution for an extended period of time determined by various qualitative assessments
* To monitor for changes in plasma levels of Cannabidiol Oral Solution during long-term treatment of subjects with IS

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification, including infantile spasms
* Parent(s)/caregiver(s) fully comprehend and sign the informed consent form, understand all study procedures, and can communicate satisfactorily with the Investigator and study coordinator.

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the analysis of results
* During the Safety Treatment and Follow-up Periods, subjects are not to receive the following:

  1. any cannabinoids (CBD, Δ9-tetrahydrocannabinol (THC), hemp oil, Realm Oil or marijuana)
  2. any other investigational drug or investigational device

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc
Locations (4):
- United States (4):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Miami Children's Hospital, Miami, Florida
  - Beaumont Health System, Royal Oak, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Months] | 23.0 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Who Are Considered Complete Responders at Day 14
Description: Complete response was defined as complete resolution of spasms and hypsarrythmia (if present at baseline) confirmed by video-electroencephalogram (EEG) at Day 14.
Time Frame: Day 14
Population: Efficacy Analysis Population: included all participants who received study drug for at least 14 days and underwent video EEG on Day 14.
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Percentage of participants | 14.3

2. Primary Outcome: Part B: Percentage of Participants Experiencing Adverse Events (AEs), Treatment-Emergent AEs (TEAEs), and Serious Adverse Events (SAEs)
Time Frame: Up to Week 64
Population: Safety Analysis Population: included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 9
Percentage of participants
  AEs | 44.4
  TEAEs | 33.3
  SAEs | 0.0

3. Secondary Outcome: Part A: Percentage of Participants With Absence of Infantile Spasms at Day 14
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Percentage of participants | 42.9

4. Secondary Outcome: Part A: Percentage of Participants With Absence of Hypsarrhythmia at Day 14
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Percentage of participants | 42.9

5. Secondary Outcome: Part A: Median Reduction in Seizure-burden Comparing Video-EEG at Baseline to Repeat Video-EEG at Day 14
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Number of spasms
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Number of spasms
  Visit 1(Baseline) | 0.0 [0 to 3]
  Visit 3 (Day 14) | 9.0 [8 to 10]

6. Secondary Outcome: Part A: Parent Impression of Efficacy and Tolerability of Study Drug
Description: Parent impression of efficacy and tolerability, as measured by Clinical Global Impression-Global Improvement Scale (CGI-I), was summarized by visit and status of response (Complete/Partial and No Response) at Visit 3 (Day 14), Visit 4 (Week 4), Visit 5 (Week 8), Visit 6 (Week 10), and end of study. The CGI-I was also analyzed in a continuous scale, as follows: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, and 7 = Very much worse
Time Frame: Visit 3 (Day 14), Visit 4 (Week 4), Visit 5 (Week 8), Visit 6 (Week 10), and end of study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Units on a scale
  Visit 3 (Day 14) | 3.0 (1.0)
  Visit 4 (Week 4): number analyzed (Participants) | 1
  Visit 4 (Week 4) | 1.0 (NA) — Only one participant was analyzed, therefore there is no standard deviation.
  Visit 5 (Week 8): number analyzed (Participants) | 1
  Visit 5 (Week 8) | 1.0 (NA) — Only one participant was analyzed, therefore there is no standard deviation.
  Visit 6 (Week 10): number analyzed (Participants) | 1
  Visit 6 (Week 10) | 1.0 (NA) — Only one participant was analyzed, therefore there is no standard deviation.
  Early Discontinuation/ End of Study: number analyzed (Participants) | 1
  Early Discontinuation/ End of Study | 4.0 (NA) — Only one participant was analyzed, therefore there is no standard deviation.

7. Secondary Outcome: Part A: Percentage of Participants With a Partial Response to Treatment
Description: Partial response was defined as a substantive change in background EEG or reduction in spasms on video EEG obtained at Day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 7
Percentage of participants | 0

8. Secondary Outcome: Part A: Percentage of Complete Responders With Relapse
Description: Complete response was defined as complete resolution of spasms and hypsarrythmia (if present at baseline) confirmed by video-EEG at Day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 1
Percentage of participants | 0

9. Secondary Outcome: Part A: Time to Complete Responder Relapse
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Days
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 1
Days | NA — No complete responders experienced relapse, therefore time to complete responder relapse could not be reported.

10. Secondary Outcome: Part B: Parent Impression of Efficacy and Tolerability of Study Drug as Measured by the Change in Clinical Global Impression of Improvement Assessment (CGI-I), Responses at Every Visit Throughout Part B
Time Frame: Up to Week 64
Population: Due to concerns of participant confidentiality this outcome measure was not analyzed. Only 1 participant participated in Part B due to study termination.
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 0

11. Secondary Outcome: Part B: Investigator Impression of Efficacy and Tolerability of Study Drug as Measured by the Change in CGI-I Responses at Every Visit Throughout Part B
Time Frame: Up to Week 64
Population: as for outcome 10
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 0

12. Secondary Outcome: Part B: Median Reduction in Seizure-burden Comparing Seizure Diaries Throughout Part B.
Time Frame: Up to Week 64
Population: as for outcome 10
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 0

13. Secondary Outcome: Part B: Percentage of Participants Who Have a Relapse of Spasms Based on Video-EEG
Time Frame: Up to Week 64
Population: as for outcome 10
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 0

14. Secondary Outcome: Part B: Time to Relapse as Confirmed by Video-EEG
Time Frame: Up to Week 64
Population: as for outcome 10
Arm/Group | Cannabidiol Oral Solution: 20 or 40 mg/kg/Day BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 64 weeks.
Groups:
- Cannabidiol Oral Solution: 20-40 mg/kg/Day BID: The dose of Cannabidiol Oral Solution will begin at 20 mg/kg/day [10 mg/kg twice per day (BID)], will be adjusted at any time if the investigator feels the safety or well-being of the participant is at risk, and will be titrated up or down according to protocol-stipulated parameters and at the investigator's discretion after Day 14 to enhance efficacy. Dose will not exceed 40 mg/kg/day.
Arm/Group | Cannabidiol Oral Solution: 20-40 mg/kg/Day BID
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol Oral Solution: 20-40 mg/kg/Day BID (N=9)
Infantile Spasms (Nervous system disorders) | 3
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Irritability (Psychiatric disorders) | 1
Sedation (Nervous system disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No